CLINICAL TRIAL: NCT06239636
Title: First-in-human Safety Study of Hypoimmune Pancreatic Islet Transplantation in Adult Subjects With Type 1 Diabetes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Per-Ola Carlsson (Other)
Collaborators: Sana Biotechnology (Industry)
Responsible Party: Sponsor-Investigator, Per-Ola Carlsson, Professor, Senior consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP421-ET1D; 2023-507988-19-00 (Other: EU CT number)
Record Dates: First submitted 2024-01-22; First posted 2024-02-02 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UP421 transplantation (Experimental): Intramuscular transplantation of study product UP421
  Interventions: Biological: UP421

INTERVENTIONS:
Biological: UP421 — Intramuscular transplantation with the ATMP UP421 composed of genetically modified human pancreatic islet cells

SUMMARY:
The current study tests the hypothesis whether genetically modified Langerhans islet cells containing insulin-producing cells from a deceased organ donor can

1. be transplanted safely and
2. help to regain insulin production in individuals with type 1 diabetes without need in simultaneous treatment with immunosuppressive medicines.

The study is an open, one-armed study where adult subjects with longstanding type 1 diabetes will receive transplantation of Langerhans islet cells (25 000 000-80 000 000) into forearm muscle. Both subjects receive active treatment. Safety is monitored with frquent follow-up visits over a year, including medical examinations, blood tests and MRI scans. Insluin producing cell function is monitored with blood samples and continuous glucose measurement.

Main objective is to to investigate the safety of an intramuscular transplantation of genetically modified allogeneic human islets (study product UP421) in adult subjects diagnosed with type 1 diabetes.

Secondary objectives are to study changes in beta-cell function, metabolic control and immunological response to pancreatic islets during the first year following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent for participation in the study
2. Diagnosis of type 1 diabetes mellitus (T1D);

   i) for ≥ 5 years and

   ii) diagnosed before the age of 18 years and

   iii) at least one or more HbA1c documented in the subject's medical journal or Swedish National Diabetes Registry during the last five-year period must be

   ≥70 mmol/mol.
3. The subject must be involved in intensive diabetes management defined as self-monitoring of subcutaneous glucose level by continuous glucose monitoring or by

   intermittent scanning glucose monitoring no less than a mean of three times per day averaged over each week and by the administration of three or more insulin

   injections per day or insulin pump therapy. This management must be under the direction of an M.D specialized in endocrinology and diabetology with support of

   a diabetes nurse at a specialist clinic for Endocrinology and Diabetology or Internal Medicine during the 12 months prior to study enrolment.
4. C-peptide negative (C-peptide < 0.01 nmol/l) in response to a mixed meal tolerance test (MMTT)
5. Positive for antibodies to either GAD or IA2 at screening
6. 30-45 years of age at time of enrollment
7. HbA1c ≥70 mmol/mol
8. Exogenous insulin needs < 1 IU/kg
9. Body weight <80 kg
10. Female subjects of child-bearing potential must agree to using adequate contraception until one year after the administration of UP421, as outlined in

https://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf

A woman is considered of childbearing potential if she is not surgically sterile or isles than 1 year since last menstrual period.

Adequate contraception is as follows:

1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal)
2. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable)
3. intrauterine device (IUD)
4. intrauterine hormone-releasing system (IUS)
5. bilateral tubal occlusion f) vasectomised partner g) sexual abstinence Male subjects must not intend to procreate until one year after the administration of UP241.

   Males must be willing to use effective measures of contraception (condoms) during the whole trial period.

   Exclusion Criteria:

   Any previous organ transplantation;

   2. Any systemic immunosuppressive medication for any other disease;

   3. Any history of malignancy;

   4. Use of any investigational agent(s) within 4 weeks of enrollment;

   5. Use of any anti-diabetic medication, other than insulin, within 4 weeks of enrollment;

   6. Active infections including Tuberculosis, HIV, HBV and HCV;

   7. Liver function test value for AST, ALT, GGT or ALP exceeding the respective reference interval for the clinical assay at Uppsala university hospital;

   8. Serological evidence of infection with HTLVI or HTLVII;

   9. Pregnancy, nursing, intention for pregnancy;

   10. Chronic kidney disease grade 3 or worse (GFR<60 ml/min as estimated by creatine measurement) ;

   11. Medical history of cardiac disease, or symptoms at screening consistent with cardiac disease;

   12. HLA immunization;

   13. MIC A/B immunization;

   14. Known autoimmune disease other than type I diabetes (e.g. Hashimoto disease);

   15. Administration of live attenuated vaccines <6 months before transplant;

   16. Islet antibodies where GADA >2000 IE/ml or IA2A >4000 IE/ml, or positive for ZnT8 auto-antibodies;

   17. Untreated proliferative diabetic retinopathy;

   18. Major ongoing psychiatric illness which the Principal Investigator judges increases the risk of noncompliance or does not allow safe participation in the study;

   19. Ongoing substance abuse, drug or alcohol; or recent history of treatment noncompliance;

   20. Known hypersensitivity to ciprofloxacin, gentamicin, or amphotericin (since these are used in the manufacturing process of UP421);

   21. Any other condition that in the opinion of the Principal Investigator does not allow safe participation in the study.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of treatment related adverse events accoridng to CTCAE v 5.0 | 12 months
  Number of treatment related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Immune evasion of implanted cells, as evaluated in systemic peripheral blood. | 12 months
  Assessed at 0 (before tx), 2, 4, 8, 12, 18, 26 and 52 weeks post-transplantation
Presence of peak C-peptide >0.01 nmol/l in response to a mixed meal tolerance test | 12 months
  Assessed at 4, 8, 12, 18, 26 and 52 weeks post-transplantation
Presence of non-fasting C-peptide concentrations >0.01 nmol/l. | 12 months
  Assessed at 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 52 weeks post-transplantation
Presence of peak C-peptide >0.20 nmol/l in response to a mixed meal tolerance test | 12 months
  Assessed at 4, 8, 12, 26 and 52 weeks post-transplantation
Survival of implanted cells as assessed by Magnetic resonance imaging | 12 months
  Assessed within 48 h after transplantation and 2, 4, 6, 8, 12, 26 and 52 weeks post-transplantation
C-peptide AUC in response to a mixed meal tolerance test | 12 months
  Assessed at 4, 8, 12, 18, 26 and 52 weeks post-transplantation
Delta changes in insulin requirement/kg BW | 12 months
  Assessed at 1, 2, 3, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 and 52 weeks transplantation when compared to before transplantation
Delta changes in HbA1c | 12 months
  Assessed at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 26 and 52 weeks post-transplantation when compared to before transplantation
Delta changes in glucose variability derived from a continuous glucose monitoring system | 12 months
  Assessed at 4, 8, 12, 18, 26 and 52 weeks post-transplantation when compared to before transplantation
Score in diabetes treatment satisfaction questionnaire | 12 months
  Assesssed at 4, 8, 12, 18, 26 and 52 weeks post-transplantation when compared to before transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Per-Ola Carlsson, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

REFERENCES:
- [Derived] Carlsson PO, Hu X, Scholz H, Ingvast S, Lundgren T, Scholz T, Eriksson O, Liss P, Yu D, Deuse T, Korsgren O, Schrepfer S. Survival of Transplanted Allogeneic Beta Cells with No Immunosuppression. N Engl J Med. 2025 Sep 4;393(9):887-894. doi: 10.1056/NEJMoa2503822. Epub 2025 Aug 4. PMID 40757665